CLINICAL TRIAL: NCT04595136
Title: A Two-arm Randomized Double-blind Study With COVID19-0001-USR Administered Via Nebulization to Patients With Mild and/or Moderate Severe Acute Respiratory Syndrome (SARS-COV-2) Infection to Decrease Viral Load
Brief Title: Study to Evaluate the Efficacy of COVID19-0001-USR in Patients With Mild/or Moderate COVID-19 Infection in Outpatient
Acronym: COVID-19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: United Medical Specialties (Other)
Responsible Party: Principal Investigator, JUAN J JALLER-RAD, Principal Investigator, United Medical Specialties
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COVID19-0001-USR
Record Dates: First submitted 2020-10-15; First posted 2020-10-20 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: SARS-CoV-2 Infection
Keywords: Coronavirus Infections; COVID-19; SARS-COV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Interventional study, randomized controlled, double-blind (i.e., active and passive control), 1 intervention group with investigative medicine, and a control group that will receive placebo intervention.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The mapping sequence will be hidden from the researcher by enrolling and evaluating participants in sequentially numbered, sealed, and stapled envelopes. To avoid the subversion of the allocation sequence, the name and date of birth of the participant will be written in the envelope, a second researcher verifies the process. The corresponding envelopes will be opened only after the enrolled participants complete all the reference assessments and assignment of the intervention by the protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COVID19-0001-USR (Experimental): Group 1 Patients with SARS-COV-2 (COVID19) positive test will receive Investigational Drug administer by nebulization ( COVID-19-0001-USR) Dosage: 3ml Frequency and Duration: Three times a day for 7 days
  Interventions: Drug: Drug COVID19-0001-USR
- Normal Saline (Placebo Comparator): Group 2 of patients with positive tests intervention SARS-COV-2 (COVID19) with placebo (i.e., normal saline 0.9% NS) plus standard baseline treatment for covid provided by Primary care provider ( Azithromycin, dexamethasone, and/or anticoagulants) Dosage: 3ml Frequency and Duration: Three times a day for 7 days
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Drug COVID19-0001-USR — COVID19-0001-USR by nebulization for patients with mild and/or moderate SARS- COV-2
  Other Names: Nebulized
  Arms: COVID19-0001-USR
Drug: normal saline — 0.9% NS via nebulization
  Other Names: 0.9% NS
  Arms: Normal Saline

SUMMARY:
Determine the efficacy and safety of COVID19-0001-USR in the treatment of SARS-COV-2 infection in mild to moderate manifestations administered via nebulization/inhalation.

DETAILED DESCRIPTION:
This is an interventional, randomized controlled, double-blind study (i.e., active and passive control), 1 intervention group will be randomized with COVID 19-001-USR, and a control group to receive a placebo intervention to assess efficacy, tolerance, and decrease viral load and clinical manifestation on patients infected with SARS-COV-2. This will be a self-administered study drug 3 times a day for 7 days

ELIGIBILITY:
Inclusion Criteria:

* Provide written consent before being included in the essay.
* Positive cases of COVID-19 (based on polymerase chain reaction or positive antigen test for SARS-CoV-2),
* Being diagnosed with mild to moderate SARS-COV-2 disease (COVID19)
* Symptomatic or asymptomatic patient, with good clinical appearance, Sat O2 at rest > 94% with room air, and without desaturation with ambulation, and without tachypnea,
* Respiratory rate < 20.
* Suspected cases of COVID-19, based on 3 criteria:

  * Fever > 38 Degrees Celsius
  * O2 saturation ≤94
* Abnormal laboratory indicators, any of them:

  * Lymphopenia <1500 cells/m3
  * C reactive protein >2 mg/L
  * Ferritin >300g/L

Exclusion Criteria:

* Existing decompensated conditions such as Diabetes Mellitus, Hypertension, Coronary Insufficiency, Coronary Artery Disease, Chronic Obstructive Pulmonary Disease (or any chronic or severe lung disease), Chronic Kidney Disease, Cancer, Immunosuppression, Mood Change
* Respiratory Frequency > 20 / min, Pulse > 120 bpm, systolic < 90 mmHg, diastolic < 60 mmHg
* The patient seems toxic and distressed, or, O2 at rest <93% in ambient air, or desaturation when ambulating
* Being diagnosed with severe SARS-COV-2 disease (COVID19)
* Patients with low oxygen saturation levels, need for ICU entry, need or likelihood of invasive mechanical ventilation
* Patients requiring bronchodilator treatment
* Patients with a known history of asthma and/or lung disease
* Patients with severe decompensated Chronic Obstructive Pulmonary Disease
* Patients who are unable to give consent or who are unable to follow up on the test group will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Change on viral load results from baseline after using COVID19-0001-USR via nebulization | Treatment Period of 7 days
  COVID19-0001-USR 1% nebulized pathway changes viral load of SARS-COV-2 virus (COVID19) in the upper and lower airways if started during the initial phase of infection

CONTACTS AND LOCATIONS:
Overall Officials: Juan Jaller, MD, Principal Investigator — United Medical Specialties; Carlos A Riveros, MD, Study Director — United Medical Specialties
Locations (1):
- Cimedical, Barranquilla, Atlántico, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pena-Silva R, Duffull SB, Steer AC, Jaramillo-Rincon SX, Gwee A, Zhu X. Pharmacokinetic considerations on the repurposing of ivermectin for treatment of COVID-19. Br J Clin Pharmacol. 2021 Mar;87(3):1589-1590. doi: 10.1111/bcp.14476. Epub 2020 Jul 17. No abstract available. PMID 32779815
- [Background] Chan JF, Yip CC, To KK, Tang TH, Wong SC, Leung KH, Fung AY, Ng AC, Zou Z, Tsoi HW, Choi GK, Tam AR, Cheng VC, Chan KH, Tsang OT, Yuen KY. Improved Molecular Diagnosis of COVID-19 by the Novel, Highly Sensitive and Specific COVID-19-RdRp/Hel Real-Time Reverse Transcription-PCR Assay Validated In Vitro and with Clinical Specimens. J Clin Microbiol. 2020 Apr 23;58(5):e00310-20. doi: 10.1128/JCM.00310-20. Print 2020 Apr 23. PMID 32132196
- [Background] Zou L, Ruan F, Huang M, Liang L, Huang H, Hong Z, Yu J, Kang M, Song Y, Xia J, Guo Q, Song T, He J, Yen HL, Peiris M, Wu J. SARS-CoV-2 Viral Load in Upper Respiratory Specimens of Infected Patients. N Engl J Med. 2020 Mar 19;382(12):1177-1179. doi: 10.1056/NEJMc2001737. Epub 2020 Feb 19. No abstract available. PMID 32074444
- [Background] Zheng S, Fan J, Yu F, Feng B, Lou B, Zou Q, Xie G, Lin S, Wang R, Yang X, Chen W, Wang Q, Zhang D, Liu Y, Gong R, Ma Z, Lu S, Xiao Y, Gu Y, Zhang J, Yao H, Xu K, Lu X, Wei G, Zhou J, Fang Q, Cai H, Qiu Y, Sheng J, Chen Y, Liang T. Viral load dynamics and disease severity in patients infected with SARS-CoV-2 in Zhejiang province, China, January-March 2020: retrospective cohort study. BMJ. 2020 Apr 21;369:m1443. doi: 10.1136/bmj.m1443. PMID 32317267
- [Background] Mitja O, Clotet B. Use of antiviral drugs to reduce COVID-19 transmission. Lancet Glob Health. 2020 May;8(5):e639-e640. doi: 10.1016/S2214-109X(20)30114-5. Epub 2020 Mar 19. No abstract available. PMID 32199468
- [Background] Zhao J, Yuan Q, Wang H, Liu W, Liao X, Su Y, Wang X, Yuan J, Li T, Li J, Qian S, Hong C, Wang F, Liu Y, Wang Z, He Q, Li Z, He B, Zhang T, Fu Y, Ge S, Liu L, Zhang J, Xia N, Zhang Z. Antibody Responses to SARS-CoV-2 in Patients With Novel Coronavirus Disease 2019. Clin Infect Dis. 2020 Nov 19;71(16):2027-2034. doi: 10.1093/cid/ciaa344. PMID 32221519
- [Background] Wagstaff KM, Sivakumaran H, Heaton SM, Harrich D, Jans DA. Ivermectin is a specific inhibitor of importin alpha/beta-mediated nuclear import able to inhibit replication of HIV-1 and dengue virus. Biochem J. 2012 May 1;443(3):851-6. doi: 10.1042/BJ20120150. PMID 22417684
- [Background] Mastrangelo E, Pezzullo M, De Burghgraeve T, Kaptein S, Pastorino B, Dallmeier K, de Lamballerie X, Neyts J, Hanson AM, Frick DN, Bolognesi M, Milani M. Ivermectin is a potent inhibitor of flavivirus replication specifically targeting NS3 helicase activity: new prospects for an old drug. J Antimicrob Chemother. 2012 Aug;67(8):1884-94. doi: 10.1093/jac/dks147. Epub 2012 Apr 25. PMID 22535622
- [Background] Yang SNY, Atkinson SC, Wang C, Lee A, Bogoyevitch MA, Borg NA, Jans DA. The broad spectrum antiviral ivermectin targets the host nuclear transport importin alpha/beta1 heterodimer. Antiviral Res. 2020 May;177:104760. doi: 10.1016/j.antiviral.2020.104760. Epub 2020 Mar 3. PMID 32135219
- See also: Nebulized ivermectin for COVID-19 and other respiratory diseases, a proof of concept, dose-ranging study in rats — https://www.researchsquare.com/article/rs-64501/v1